CLINICAL TRIAL: NCT03935269
Title: Can We Relieve the Stress: Cereset for Caregivers
Brief Title: Cereset for Caregivers
Acronym: CERESET
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accruals, DSMB/PRC closed study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00058097; CCCWFU 03618 (Other: Wake Forest Baptist Comprehensive Cancer Center); NCI-2019-02840 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2019-04-25; First posted 2019-05-02 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Glioma
Keywords: High-grade glioma; Stress; Caregivers
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention with Ambulatory Therapy (Experimental): Caregivers of participants with high-grade glioma will undergo standard Cereset Research Office (CRO) in-office treatment for a total of five (5) treatments. Ambulatory therapy with the Cereset Research Wearable (CRW) will be available to caregivers while they are attending routine radiation therapy with glioma patients.
  Interventions: Device: Cereset Research Wearable; Procedure: Stress management therapy; Other: Questionnaire administration; Other: Quality of Life Assessment

INTERVENTIONS:
Device: Cereset Research Wearable — CRW is a stress-relaxation device where participants listen to sounds that help to balance brain rhythms. Participants will be asked to come to an office for 5 days over 1-2 weeks, on your their schedule. Sessions will take approximately one (1) hour to complete.
Procedure: Stress management therapy — Undergo Cereset research office intervention
Other: Questionnaire administration — Ancillary studies
Other: Quality of Life Assessment — Ancillary studies

SUMMARY:
In this single arm, open label study, investigators will evaluate the feasibility of using the Cereset (formerly known as HIRREM - high-resolution relational, resonance-based electroencephalic mirroring) intervention for a stressed population confronting an acute burden on their lives - caregivers of newly diagnosed high-grade glioma patients. The Cereset intervention is a closed-loop acoustic stimulation intervention that has been studied in patients with PTSD, insomnia, postural orthostatic tachycardia, and military veterans.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the feasibility of completing the prescribed Cereset Research Office intervention for trial participants in this single arm, open label study.

Secondary Objectives

* To assess the tolerability of the intervention
* To assess changes in trial participant wellbeing and quality of life.
* To assess changes in physiological response at pre-intervention and post-intervention time points.

Exploratory Objectives

* To assess the utilization of Cereset Research Wearable (portable, limited scope wearable device) after the CRO intervention.
* To assess the participant acceptability of the Cereset Research Intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Identified as caregiver by patient with glioma as defined as the primary, non-professional, non-paid person who provides the majority of emotional financial and/or physical support. There will only be one trial participant allowed per patient/caregiver dyad.
* The trial participant must be caring for a patient who is:
* ≥18 years of age
* Has a histologically confirmed malignancy that is a high grade glioma which includes (astrocytoma, oligodendroglioma, glioblastoma, ependymoma).
* Any World Health Organization (WHO) grade gliomas
* Trial participant is able to understand and the willingness to sign an IRB-approved informed consent document.
* Trial participant is able to sit in a chair for 90 minutes.

Exclusion Criteria:

* Trial participant is a heavy alcohol user per the Substance Abuse and Mental Health Services Administration.

  * Heavy alcohol use is defined as binge drinking on 5 or more days in the past month.
  * Binge drinking is defined as 4 drinks for women and 5 drinks for men on the same occasion.
* Trial participant has severe hearing impairment defined as word discrimination at <50% with or without the use of hearing aids.
* Trial participant's weight is greater than or equal to 400 pounds at time of enrollment (chair limit).
* Prior trial participant use of transcranial magnetic stimulation (TMS), transcranial direct current stimulation (TDCS), alpha stimulation, neurofeedback, biofeedback, or deep brain stimulation (DBS) within one month before enrollment.
* Trial participant has previously used HIRREM, or Cereset.
* Trial participant has a known seizure disorder requiring ongoing anti-epileptics prescribed specifically for seizure disorder.
* Trial participant states he or she will not be able to abstain from daily use of alcohol or recreational drugs during the intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of Completed Interventions | 10 days
  Intervention feasibility will be the number of trial participants who complete the Cereset Research Office intervention (5 out of 5 prescribed sessions).

SECONDARY OUTCOMES:
Incidence of Adverse Events During Cereset Research Office Intervention | 4 months
  Tolerability will be reported as the total number, grade, time from enrollment and time to resolution of CTCAE and adverse event detected by investigator monitoring and assessment of adverse events at visits 1, 2, 3, and 4 during Cereset Research Office Intervention using the CTCAE 5.0 (Grade 1-5, 1 = mild, 5 = death). Adverse events will be divided into four categories (common adverse events >15-20%, uncommon adverse events <15%, rare but potentially serious adverse events and unexpected toxicities). Any Grade 3 toxicity by CTCAE will be further evaluated as an unacceptable event.
Caregiver Interview | 4 months
  Caregiver interview is a 21-item questionnaire that contains things a person might do when caring for a loved one with cancer. Scores ranges from 1-9 ('1' would state that the participant is not-at-all confident to accomplish the listed behavior; '9' would state that the participant is totally confident to accomplish the listed behavior. Numbers in the middle of the scale indicate that the participant is moderately confident to accomplish the listed behavior). Mean core values for each survey will be calculated for all participants enrolled. Surveys will be provided to participants pre- and post-intervention. Paired student's t-test will be used to compare scores at these V1, V2, V3, V4 time points.
Generalized Anxiety Disorder 7-item scale (GAD-7) | 4 months
  The Generalized Anxiety Disorder-7 is a validated, short seven item scale. Response scale = (not at all sure = 0; several days = 1; over half the days = 2; to nearly every day = 3). Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. Mean core values for each survey will be calculated for all participants enrolled. Surveys will be provided to participants pre- and post-intervention. Paired student's t-test will be used to compare scores at these V1, V2, V3, V4 time points
Insomnia Severity Index (ISI) | 4 months
  The Insomnia Severity Index is a validated, 7 item self-report questionnaire assessing the nature, severity, and impact of insomnia in the past month. Rating scale (0 = very satisfied to 4 = very dissatisfied; 0 = not at all noticeable to 4 = very much noticeable; 0 = not at all worried to 4 = very much worried; 0 = not at all interfering to 4 = very much interfering). Mean core values for each survey will be calculated for all participants enrolled. Surveys will be provided to participants pre- and post-intervention. Paired student's t-test will be used to compare scores at these V1, V2, V3, V4 time points
Perceived Stress Scale Questionnaire | 4 months
  The Perceived Stress Scale (PSS) is a 10-item psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Scale range is 0 = never, 4 = very often. Mean core values for each survey will be calculated for all participants enrolled. Surveys will be provided to participants pre- and post-intervention. Paired student's t-test will be used to compare scores at these V1, V2, V3, V4 time points
Changes in Heart Rate - FAROS 180 device | 4 months
  Continuous readings of heart rate will be acquired using FAROS 180 heart rate monitor for a minimum of 10 minutes for physiologic changes in heart rate at pre-intervention (B1) and during, and post-intervention time points (B2, B3, B4). The mean values of HRV will be compared with paired student's t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No